CLINICAL TRIAL: NCT06290635
Title: Edmonton Dyspnea Inventory (EDI) in Interstitial Lung Diseases: Understanding Dyspnea Severity and Impact of EDI Use in Individuals With Interstitial Lung Disease
Brief Title: Edmonton Dyspnea Inventory- Validation Study
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00119668
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: ILD
Keywords: ILD, Dyspnea, symptoms
MeSH Terms: conditions — Lung Diseases, Interstitial; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants include IPF and F-ILD including progressive pulmonary fibrosis phenotype
  Interventions: Diagnostic Test: Breathlessness Assessment Tool

INTERVENTIONS:
Diagnostic Test: Breathlessness Assessment Tool — Participants will complete a breathlessness assessment tool (questionnaire) at three timepoints over the study duration, among other validated questionnaires.

SUMMARY:
Breathlessness is a common problem for many patients with Interstitial lung disease (ILD). ILD is a group of lung diseases that cause inflammation (swelling) and scarring in the lung tissue where gas exchange (oxygen and carbon dioxide) occurs. Unfortunately, there is no cure for these conditions and as a result many patients decline over time with worsening breathlessness. This limits their ability to live a good life. Clinicians do not often recognize, assess, or treat breathlessness appropriately. Breathlessness, being a subjective experience, cannot be fully understood through objective measurements such as lung function tests, the arterial blood gas test etc. The objective and subjective measures of breathlessness are frequently disconnected. Clinicians who often rely on these types of objective tests do not directly enquire into its nature and severity of breathlessness from patients themselves. As a result, they remain unaware of this disabling symptom and the extent of its impact on patients. While there are many tools to measure breathlessness, they are not consistently used in routine care or have impacted care in a meaningful way. Many such tools are also complex with intricate response systems with possibility of errors and user fatigue. As a result, easy to use tools like modified MRC or MRC are frequently used even though they do not assess severity of breathlessness. No tool has been effective at helping clinicians identify the problem and prescribe appropriate treatments. This results in needless suffering for patients and their families and prevents them from receiving timely and appropriate therapies. Investigators propose to test an easy-to-use tool that combines the subjective and objective aspects of breathlessness. Investigators hope that the tool will help clinicians quickly identify the patient's breathlessness severity and provide them with an algorithm of what to do next. The tool was developed by clinicians with +15 years of experience in ILD and dyspnea. Early analysis already suggests the tool is useful to patients and helps improve care.

DETAILED DESCRIPTION:
Dyspnea or breathlessness is a disabling and distressing symptom that affects every aspect of a patient and caregiver's life. It is prevalent in progressive pulmonary fibrosis (PPF) as well as many other fibrotic ILD (F-ILD). Idiopathic pulmonary fibrosis (IPF), the most common and well-studied F-ILD with a life expectancy of only 3-4 years, has a dyspnea prevalence of 90% at diagnosis. Despite the high dyspnea burden in IPF and PPF and its' impact on both health-related quality of life (HRQOL) and mortality, healthcare professionals often do not adequately assess or treat dyspnea in practice. Many reasons have been proposed for this care gap.

Dyspnea is a subjective and complex symptom where experience is shaped by a variety of factors, including physiological, psychological, and environmental influences. Degree of lung function impairment does not consistently predict level of breathlessness and cannot be used as a surrogate for direct dyspnea measures. Unfortunately, dyspnea is not frequently assessed in care. Many scales exist including uni- and multidimensional scales. MRC, a unidimensional scale, is the most commonly used dyspnea scale. The MRC scale assesses dyspnea by asking which activities, ranging from vigorous exercise to minimal activities of daily living, are limited by dyspnea. The MRC scale has shown good utility in many studies. A major drawback of the MRC scale in some populations is the lack of a scale point for patients who experience dyspnea at rest, but it is easy to extend the scale to ask about dyspnea at rest. However, scales such as the MRC are indirect; they do not actually ask the patient how much dyspnea they experience. Experts have therefore recommended that patients not only be routinely asked about dyspnea but should also be asked to rate its severity. In a recent study of over 67000 patients, dyspnea severity reported by patients during a rapid nursing assessment on admission was associated with two-fold odds of death in 2 years. The authors noted that patients who reported any dyspnea were at an increased risk of death during that hospital stay, the greater the dyspnea severity, the greater the risk of death. Even after adjustment for patient comorbidities, demographics, and severity of illness, increasing dyspnea severity remained associated with inpatient mortality. They suggest that routine assessment of dyspnea severity may allow for better monitoring and optimal interventions that could potentially reduce mortality and morbidity. A 2015 survey of US-based hospitalists also suggests that dyspnea severity may help guide management. Unfortunately, routine dyspnea severity assessment is also uncommon in practice.

Secondly there are no dyspnea treatment algorithms for clinicians to implement in practice. The American Thoracic Society (ATS) statements and guidelines emphasize the urgent need to assess and manage dyspnea in respiratory disease, including IPF but do not provide a treatment algorithm. They do recommend evidence-based therapies such as pulmonary rehabilitation, anxiolytics and opioids and the treatment of associated psychosocial factors. And finally, physician perspectives regarding dyspnea and reluctance to use opiates, inadequate education and lack of training are all important barriers to effective dyspnea management.

To address this care gap in assessment, investigator developed an easy-to-use scale, Edmonton Dyspnea Inventory (EDI) in the Multidisciplinary Collaborative ILD Clinic, Edmonton, Canada. EDI is a pilot tool to assess dyspnea severity at rest, during activities of daily living and self-reported exercise. In addition, the tool also documents crisis dyspnea episodes and their triggers to guide management. Investigator's preliminary work showed that EDI has good internal consistency, strong correlation with MRC and weak correlation with lung function data. Group based trajectory modelling showed 3 different groups of dyspnea intensity with implications for survival. Investigator also showed feasibility of outpatient clinical use over 10 years. In addition, EDI use led to early institution of dyspnea therapies (van Den Bosch AJHPC 2023). This tool facilitated early and personalized dyspnea management that differs both between and within individual MRC grades (Kalluri. AJHPC 2024). Investigator has also shown this approach to dyspnea assessment and management facilitates patient self-management and mastery, allowing reduction in acute care utilization and healthcare costs in IPF. This is the only tool to that facilitates both assessment and management of dyspnea. Systematic assessment and appropriate dyspnea management is an urgent unmet need in patient care. Physicians and clinicians require an easy-to-use tool to assess dyspnea and create a personalized management plan for their patients. Investigator believes EDI can serve both purposes as per our early studies. Investigator proposes to examine EDI's cross-sectional and longitudinal validity and reliability for use in IPF and F-ILD including PPF. Investigator will also explore patient and care provider perceptions on the use of EDI and its potential/actual impact on clinical care using focus group methodology. Investigator will recruit participants from all three sites for qualitative analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a guideline-based diagnosis of IPF and any fibrotic ILD including progressive pulmonary fibrosis (PPR).
* All adult patients with the condition of interest will be recruited regardless of age, gender, ethnicity, stage of disease to enable broad inclusion.
* As IPF is male dominant disease with most cases presenting late, we need to ensure that females and milder dyspnea grades (MRC 1-2) are also represented in the sample. Dyspnea perception is expected to be higher in females. To ensure representative sampling, we will use a sampling frame at 50% enrolment (50 patients) to ensure at least 25% females and smaller dyspnea grade are included at that point. If not, recruitment will be modified to achieve this.

Exclusion Criteria:

* Participants unable to consent or understand English or Danish will be excluded as we do not have a version of the scale translated in other languages.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ILD patients with age > 18 yrs with diagnosis confirmed by ILD experts and included IPF, PPF or F-ILD
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Validate Edmonton Dyspnea Inventory (EDI; formerly known as multidimensional dyspnea scale-MDDS) | 6 months
  Several validity and reliability analyses will be conducted in a cohort of IPF and F-ILD patients (concurrent or face validity); Scale consists of 9 questions that yield a total score between 0-90 with higher scores indicating worse breathlessness

SECONDARY OUTCOMES:
To perform time-motion observation of care providers or patients using the scale | 1
  To perform time-motion observation of care providers or patients using the scale
Calculate MCID for Edmonton Dyspnea Inventory | 6 months
  To Calculate minimum clinically important difference in Edmonton Dyspnea Inventory scores between baseline and 6 months follow up. Scale consists of 9 questions that yield a total score between 0-90 with higher scores indicating worse breathlessness
Feasibility of Questionnaire | 6 months
  To assess feasibility and acceptance amongst IPF and F-ILD patients and clinicians (Physicians-ILD and Palliative Care and allied health)
To assess day-to-day variability in dyspnea scores | 1 week
  We will assess variability over a few observations for 1 week follow-up period. Scale consists of 9 questions that yield a total score between 0-90 with higher scores indicating worse breathlessness

CONTACTS AND LOCATIONS:
Locations (3):
- Kaye Edmonton Clinic, Edmonton, Alberta, Canada
- Aarhus University, Aarhus, Denmark
- Bristol ILD Service; North Bristol NHS Trust, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No